CLINICAL TRIAL: NCT02239328
Title: A Study of Patient-reported Outcomes in Patients With Lung or Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Alliance for Clinical Trials in Oncology (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Benjamin Kozower, MD, Principal Investigator, University of Virginia
Other Study IDs: 17525
Record Dates: First submitted 2014-08-20; First posted 2014-09-12 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-01

CONDITIONS: Lung Cancer; Esophageal Cancer
Keywords: Lung cancer; esophageal cancer
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung Cancer, Esophageal Cancer: Lung Cancer and Esophageal Cancer patients will complete the online PROMIS survey. No treatment intervention will be performed.

SUMMARY:
This survey study is looking to determine if patient reported outcomes(using the PROMIS survey) will vary according to the presence of recurrent or metastatic lung or esophageal cancer.

DETAILED DESCRIPTION:
A patient-centered approach to lung cancer surveillance following resection needs to incorporate patient reported outcomes. The Patient Reported Outcomes Measurement Information System (PROMIS®) was designed to revolutionize the assessment of patient reported outcomes by establishing a national resource for the measurement of patient-reported symptoms and other health outcomes.

The PROMIS Assessment Center, the management tool within the larger PROMIS system, will be used to securely store de identified data, provide automated accrual reports and data export for this specific study. This study will have it's own study specific website.

Patients seen at the University of Virginia Cancer Center will be identified and invited to participate in an assessment of their reported outcomes over multiple domains available in PROMIS. Collecting this information on lung cancer survivors may provide a robust platform to design a patient-centered surveillance strategy following resection.

The study team hypothesizes that patient reported outcomes will vary according to the presence of recurrence or metastasis of lung or esophageal cancer. The study team also believes including patient reported outcomes into routine post-treatment surveillance will improve patient satisfaction and improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Suspected or Known diagnosis of lung or esophageal cancer
* Willing and able to complete questionnaires

Exclusion Criteria:

* Subjects unwilling to provide informed consent
* Subjects unwilling or unable to answer the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer Esophageal cancer
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2014-08; Primary Completion 2017-06 (Actual); Study Completion 2017-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Kozower, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and recruited in the Thoracic surgery clinic during their appointments. Subject recruitment began on 08/20/2014 and was completed on 11/20/2015.
Pre-assignment Details: There was no wash out or run-in period for this study. Subjects were consented and then immediately completed the survey.
Period: Overall Study
Arm/Group | Lung Cancer, Esophageal Cancer
Started | 182
Completed | 174
Not Completed | 8
Not completed — Benign disease noted at time of surgery | 6
Not completed — Equipment or website malfunction | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lung Cancer, Esophageal Cancer
Number analyzed (Participants) | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92
  Male | 82
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 174
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 162
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 174
Current smokers [Count of Participants; unit: Participants] | 53

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Scores.
Description: Enrolled subjects with lung or esophageal cancer will be asked to complete an on-line (web-based) survey (PROMIS) using a computer. Most patients will only be asked to complete this survey once, but some patients will be asked to answer the questions a second or third time over a maximum five year period. The PROMIS assessment center was used to develop and administer patient reported outcomes (PROs) for each of these five cancer domains. PROMIS scores are continuous and range from 0-100. Total scores were calculated and calibrated to the weighted distribution of scores from a large representative sample of the U.S. general population using the 'T-score' algorithm 18. The T-scores for the study population are calibrated to the surveyed population mean of 50 and standard deviation of 10, such that a study patient with a T-score of 40 is one standard deviation below the U.S. general population mean.
Time Frame: Over a 3 year period
Population: All patients who completed at least 1 PROMIS survey who had a diagnosis of lung cancer.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lung Cancer, Esophageal Cancer
Number analyzed (Participants) | 174
units on a scale
  Physical Function | 43.05 (8.57)
  Anxiety | 51.51 (9.27)
  Depression | 48.64 (8.68)
  Fatigue | 50.74 (9.66)
  Pain | 51.45 (9.37)
Statistical Analysis 1: Comparison: Lung Cancer, Esophageal Cancer; Test type: Other — Multilevel random coefficient models estimated the mean score of each PROMIS domain as a function of time elapsed between date of surgery and assessment (in years), and patient comorbidity. Statistical significance of estimated fixed effects were assessed by the F-test statistic for type 3 tests, p < 0.05; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Over a 3 year period
Description: An adverse event will be considered any undesirable sign, symptom or medical condition considered related to the intervention. Medical conditions/ diseases present before starting the intervention will be considered adverse events only if they worsen after starting the study and that worsening is considered to be related to the study intervention. OR any undesirable and unintended effect of research occurring in human subjects as a result of collection of private identifiable information.
Arm/Group | Lung Cancer, Esophageal Cancer
All-Cause Mortality (participants affected / at risk) | 0/174
Serious Adverse Events (participants affected / at risk) | 0/174
Other Adverse Events (participants affected / at risk) | 0/174

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-07-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT02239328/Prot_SAP_000.pdf
  • Informed Consent Form (2014-07-31): https://cdn.clinicaltrials.gov/large-docs/28/NCT02239328/ICF_001.pdf